CLINICAL TRIAL: NCT00068094
Title: The Effect of a Probiotic on Hepatic Steatosis
Brief Title: The Effect of Good Bacteria on Nonalcoholic Fatty Liver Disease in Diabetics
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001305 (NIH)
Record Dates: First submitted 2003-09-05; First posted 2003-09-09 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Fatty Liver; Hepatic Steatosis; Diabetes Mellitus; Liver Diseases
Keywords: Probiotics; Bacteria
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus; Liver Diseases

INTERVENTIONS:
Drug: Probiotic-containing powder

SUMMARY:
The purpose of this study is to determine whether probiotics, bacteria that may improve liver health, can effectively treat a chronic condition in diabetics that increases fat in the liver.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in the United States and is also common in diabetics; unfortunately, research on NAFLD has been limited. Safe, inexpensive, and well-tolerated treatments for NAFLD are needed. Recent studies indicate that probiotics help to improve fat breakdown in mice. This study will evaluate the efficacy of probiotic therapy to reduce fat accumulation in the livers of people with NAFLD and diabetes.

Participants in this study will be randomly assigned to receive either a probiotic-containing mixture or placebo once daily for 6 months. Blood tests, and magnetic resonance spectroscopy will be used to assess participants at study start and at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Nonalcoholic fatty liver disease

Exclusion Criteria:

* Any cause of liver disease other than hepatic steatosis
* Diabetes
* Known or suspected cirrhosis
* Inability or unwillingness to undergo magnetic resonance procedures
* Requirement of long-term antibiotic therapy
* Pregnancy, breast-feeding, or plans to become pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-07; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Steve Solga, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Solga SF, Diehl AM. Non-alcoholic fatty liver disease: lumen-liver interactions and possible role for probiotics. J Hepatol. 2003 May;38(5):681-7. doi: 10.1016/s0168-8278(03)00097-7. No abstract available. PMID 12713883
- [Background] Li Z, Yang S, Lin H, Huang J, Watkins PA, Moser AB, Desimone C, Song XY, Diehl AM. Probiotics and antibodies to TNF inhibit inflammatory activity and improve nonalcoholic fatty liver disease. Hepatology. 2003 Feb;37(2):343-50. doi: 10.1053/jhep.2003.50048. PMID 12540784